CLINICAL TRIAL: NCT06820892
Title: Evaluation of the Concordance Between the Information Delivered in Antenatal Diagnosis Consultation and Parents Experience After the Birth of Their Infant
Brief Title: Quality of Information Provided During Antenatal Consultations
Acronym: EVIDANCE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5216
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Congenital Anomalies; Prematurity; Antenatal Consultation
Keywords: Antenatal; Antenatal consultation; information
MeSH Terms: conditions — Congenital Abnormalities; Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients (mother only): The patients were observed in a multidisciplinary prenatal diagnosis centre and subsequently delivered a newborn infant, who was then admitted to the neonatology department of the same hospital, between January 2020 and December 2022.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The study utilised a 16-item questionnaire to evaluate the quality of information received during antenatal diagnosis consultations and its congruence with subsequent experiences following birth and hospitalisation of the infant. The questionnaire encompassed seven questions pertaining to consultation arrangements, including duration, frequency and unit visits, six questions addressing the received information, and three questions exploring the long-term outcomes of the child.

SUMMARY:
The objective of this questionnaire study is to evaluate the concordance between the information provided to parents during antenatal consultations and their subsequent experiences following childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Patients were observed at the multidisciplinary prenatal diagnosis centre.
* Patients who had attended at least one antenatal consultation with a pediatric neonatologist
* Patients who gave birth between January 2020 and December 2022 and whose newborn was hospitalized in the neonatology department

Exclusion Criteria:

* a child who died in hospital or had a condition with a high risk of death in the first few years of life
* non-French speaking mothers
* Mothers who were minors at the time of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Of the patients who were followed up at the multidisciplinary prenatal diagnosis centre and had an antenatal consultation with a pediatric neonatologist, 113 patients met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Question 8 of the questionnaire | The outcome is measured at the time of questionnaire completion, typically at hospital discharge or within one week post-discharge.
  In summary, did the information provided during the consultation with the paediatrician correspond to the events that transpired during your child's hospitalisation ? Patients are invited to indicate their level of agreement or disagreement with a series of four statements by selecting one of four options : 'not at all', 'to some extent', 'almost' or 'completely'.

CONTACTS AND LOCATIONS:
Locations (1):
- Femme Mère Enfant Hospital (HFME), Bron, France